CLINICAL TRIAL: NCT01211639
Title: Genetic Evaluation of Natalizumab-Treated Patients With Progressive Multifocal Leukoencephalopathy
Status: Terminated | Type: Observational
Why Stopped: Due to lack of enrollment.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 101JC403
Record Dates: First submitted 2010-09-16; First posted 2010-09-29 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Progressive Multifocal Leukoencephalopathy
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood collection for genetic analysis Urine collection for archiving and future research use Plasma, Serum, and Peripheral Blood Mononuclear Cells (PBMC) collection for archiving and future research use
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to explore host genetic mutations which may render individual subjects more susceptible (or resistant) to developing Progressive Multifocal Leukoencephalopathy (PML). Samples will also be collected to determine Deoxyribonucleic Acid (DNA) sequence of JC Virus (JCV). Analysis of the JC Virus (JCV) genome may provide information about viral genotypes that may be associated with higher pathogenicity, and help to identify individuals who may be at higher risk of developing Progressive Multifocal Leukoencephalopathy (PML) due to chronic infection with a more pathogenic variant of JC Virus (JCV).

DETAILED DESCRIPTION:
Deoxyribonucleic acid (DNA) will be analyzed from natalizumab-treated subjects who develop Progressive Multifocal Leukoencephalopathy (PML). The genetic analysis of the subjects will directly seek mutations that could identify subjects at risk.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects who have confirmed PML while on treatment with Natalizumab

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in subjects who have confirmed Progressive Multifocal Leukoencephalopathy (PML) while being treated with natalizumab.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
to examine host genetic variation and possible genetic susceptibility to PML | Up to 3 Months

SECONDARY OUTCOMES:
To explore predisposing factors of the innate and adaptive immune system | Up to 3 Months
To analyze DNA sequences of JCV | Up to 3 Months
optional substudy: to test alterations in DNA repair pathways | Up to 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (11):
- United States (10):
  - North Central Neurology Associates, Cullman, Alabama
  - Rocky Mountain MS Center at Anschutz Medical Campus University Colorado Denver, Aurora, Colorado
  - Rush Medical Center - Rush Multiple Sclerosis Center, Chicago, Illinois
  - St. Vincent Hospital, St. Vincent Neuroscience Institute, Indianapolis, Indiana
  - Central Neurology, Hastings, Nebraska
  - Clinical Research Center UH, The Nebraska Medical Center, Omaha, Nebraska
  - NYU Hospital for Joint Disease, MS Care Center, New York, New York
  - University of Rochester, Rochester, New York
  - Research Site, Cincinnati, Ohio
  - Neurology of Bend, LLC, Bend, Oregon
- Research Site, Würzburg, Germany